CLINICAL TRIAL: NCT06617585
Title: The Role of CircDENND4C in Epithelial Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mamdouh Mohamed Abdellah, doctor, Assiut University
Other Study IDs: CircDENND4C in ovarian cancer
Record Dates: First submitted 2023-11-27; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
circular RNAs (circRNAs), a newly discovered type of endogenous noncoding RNAs [8], are involved in the regulation of various biological functions. They act by sponging off certain microRNAs (miRNAs) and play a role in the pathogenesis of many diseases, including cancers [9-11]. In addition, circRNAs are not com- monly degraded by RNA enzymes present in body flu- ids [8], and most of them possess expression specificity at the tissue, cell, and developmental stage level [12,13]. Thus, they can be ideal clinica

DETAILED DESCRIPTION:
epithelial OC (EOC), the most common form of OC, accounts for 90% of all OC cases [2]. EOC has the highest mortality among all gynecologic tumors and poses a serious threat to women's life [3].herefore, early clinical diagnosis is crucial. Commonly used laboratory indicators for OC diagnosis

ELIGIBILITY:
Inclusion Criteria:

- patients at South Egypt Cancer institute and Recently diagnosed ovarian cancer patients 2. Patients not went to surgery.

Exclusion Criteria:

* . Patients receive any anti-cancer therapy. 2. Patients diagnosed with other concomitante cancer or chronic disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: apparently healthy group and group of known diagnosed as ovary cancer in assiut uni hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-02-02 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
role of circDENND4c in the diagnosis of ovarian cancer | baseline
  by quality real time PCR we use the circDENND4c as a tumour marker for ovarian cancer

IPD SHARING:
Plan to Share IPD: No